CLINICAL TRIAL: NCT03900910
Title: A Gastric Cancer Prevention Program for Aboriginal People Living in the Remote Areas
Brief Title: Gastric Cancer Prevention for Indigenous Peoples
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201804108RINB; 1070056368 (Other: Council of Indigenous Peoples in Taiwan)
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Gastric Cancer
Keywords: Cancer prevention; Antibiotics; Inequality
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Mass screening and eradication of Helicobacter pylori infection in Indigenous community.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastric cancer prevention (Experimental): 13C-urea breath test and anti-H. pylori treatment for those who are tested positive.
  Interventions: Other: Gastric cancer prevention; Other: Execution of the program
- The acceptability and applicability of the mass screening program (Experimental): Our short-term outcome is the acceptability and feasibility of this screening program, which will be evaluated by answering whether the screening quality indicators can reach the minimal requirements.
  Interventions: Other: Gastric cancer prevention; Other: Execution of the program

INTERVENTIONS:
Other: Gastric cancer prevention — Participants will receive the 13C-urea breath test and those with test positive will further receive H. pylori eradication treatment.
Other: Execution of the program — Screening program is audited by the standardized quality indicators, including the participation rate, the positivity rate, the referral-to-treatment rate, and the eradication rate .

SUMMARY:
The incidence of gastric cancer in local indigenous peoples is higher than the non-Indigenous counterpart in Taiwan. How to design an effective prevention strategy for gastric cancer is of importance. The present study aimed to identify the causes that may account for the health inequalities, allowing generation of a plan of action on the whole population scale.

DETAILED DESCRIPTION:
Owing to the continuing gap in cancer burden between Indigenous and non-Indigenous peoples, reducing health disparities has drawn worldwide attention. Evidence indicates that the gastric cancer incidence and mortality rates in Indigenous peoples are much higher than those of non-Indigenous counterparts living in the same areas. Exposure to more risk factors from social habits, lifestyle, and Helicobacter pylori infection has been considered the cause. However, even though gastric cancer has been repeatedly shown to be preventable by eliminating risk factors, eradication policies are rarely designed for Indigenous peoples. Possible obstacles may include the lack of Indigenous health statistics, inadequate access to care, difficulty in modifying social habits and lifestyles, and the presence of environmental and cultural barriers. Developing and implementing a preventive strategy following the evidence-based principle remains a challenge.

In Taiwan, the number of Indigenous peoples has grown; however, their life expectancy remains substantially lower than that of the non-Indigenous population. Cancer is the most prevalent cause of death for Indigenous peoples and a disproportionate prevalence of certain kinds of cancer is noted for Indigenous peoples. These observations provide an opportunity to establish a plan of action, in which a specific intervention is developed to decrease the threat from each specific cancer so that the overall disparate burden can be reduced in a stepwise manner.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-60 years
* Mentally competent to be able to understand the consent form
* Able to communicate with study staff for individuals

Exclusion Criteria:

* Pregnancy
* Individuals with major comorbid diseases

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Gastric cancer incidence | After at least 5 years, the gastric cancer incidence per 100,000 person-years is calculated by the person-years of follow-up.
  To assess the effect of H. pylori eradication for gastric cancer prevention
Helicobacter eradication rate | At least 5 years
  To assess the eradication rate of anti-H. pylori treatment.
The participation rate | Screening program quality indicator
  The number of participants divided by the number of invitees
The positivity rate | Screening program quality indicator
  The number of positive test results divided by the number of participants
The referral-to-treatment rate | Screening program quality indicator
  The number of individuals who received anti-H pylori treatment divided by the number of positive test results
The reinfection rate | Screening program quality indicator
  The number of positive test results divided by the person-years of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Chia Lee, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
No individual participant data could be shared.

REFERENCES:
- [Derived] Lei WY, Lee JY, Chuang SL, Bair MJ, Chen CL, Wu JY, Wu DC, Tien O'Donnell F, Tien HW, Chen YR, Chiang TH, Hsu YH, Hsu TH, Hsieh PC, Lin LJ, Chia SL, Wu CC, Subeq YM, Wen SH, Chang HC, Lin YW, Sun KP, Chu CH, Wu MS, Graham DY, Chen HH, Lee YC. Eradicating Helicobacter pylori via 13C-urea breath screening to prevent gastric cancer in indigenous communities: a population-based study and development of a family index-case method. Gut. 2023 Nov 24;72(12):2231-2240. doi: 10.1136/gutjnl-2023-329871. PMID 37197905
- See also: Action Plans to Reduce Health Disparity in Indigenous Communities in Taiwan — https://dep.mohw.gov.tw/DONAHC/lp-3949-104.html